CLINICAL TRIAL: NCT05246449
Title: Multi-centre, National, Randomised, Exploratory Study Evaluating the Benefit of an Individualised Treatment Plan(VitalCare) Compared to Standard of Care, in Obstructive Sleep Apnoea Patients Treated With CPAP/APAP
Brief Title: Evaluate the Benefit of an Individualised Treatment Plan (VitalCare) VS SOC in OSA Patients Treated With CPAP/APAP
Acronym: VitalCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Collaborators: Clinact (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ALMED-21-001
Record Dates: First submitted 2022-01-27; First posted 2022-02-18 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Sleep Apnoea Syndrome (OSAS)
Keywords: CPAP/APAP; VitalCare; homecare provider; individualised treatment plan
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care group (No Intervention): with patients starting their regular CPAP/APAP treatment without stratification, with medical follow-up, and with standard home CPAP/APAP service provided by home healthcare,
- VitalCare group (Experimental): with patients starting their CPAP/APAP treatment and with a personalized follow-up by the homecare provider.
  Interventions: Other: individualised treatment plan (VitalCare) and associated remote medical monitoring

INTERVENTIONS:
Other: individualised treatment plan (VitalCare) and associated remote medical monitoring — VitalCare is a treatment plan to help in the personalisation of patient care.
  Arms: VitalCare group

SUMMARY:
According to a stratification procedure, the objective of a personalised care plan (VitalCare) is to identify points for improvement since the early stage of the patient's pathway of CPAP/APAP treatment and to adjust patient follow-up .

DETAILED DESCRIPTION:
It is a prospective, exploratory, randomised, multi-centre, open, controlled study with a 1:1 ratio of two parallel groups, with obstructive sleep apnoea patients starting CPAP/APAP therapy, and receiving by the homecare provider, either an individualised treatment plan (VitalCare) or national standard of care.

This study will be conducted in 5 hospital centres in Portugal..

During a regular medical consultation, eligible patients who have signed their informed consent will be randomised by their investigator.

Two study groups will be set up:

1. Standard of care group
2. VitalCare group

Two medical visits in the hospital centres will be scheduled in the context of the study for all participating patients:

1. A screening/inclusion visit before CPAP/APAP initiation at home;
2. An end-of-study visit planned at 12 months (± 1 month) after CPAP/APAP initiation at home. All visits done in the hospital centres at the discretion of the investigators between patient's screening/inclusion visit and end-of-study visit will be recorded in the eCRF with the reason for the visit and change in CPAP/APAP prescription, if applicable

The primary objective of this study is to evaluate adherence to CPAP/APAP treatment at 3 months in patients with individualised treatment plan (VitalCare) compared to patients with standard of care

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with Obstructive Sleep Apnoea Syndrome (OSAS) who is newly prescribed CPAP or APAP therapy at inclusion
* Patient agreeing to the collection of data from their CPAP/APAP device via teletransmission
* Patient equipped with a device compatible with the ResMed telemonitoring data platform
* Patient who has signed the informed consent form for the study

Exclusion Criteria:

* Obese patient presenting hypoventilation
* Patient at risk of other sleep disorders (e.g. severe insomnia)
* Patient with physical, mental or cognitive inability to use all components of the remote medical monitoring project and individualised treatment plan, as determined by the investigator wishing to include the patient
* Patient with severe COPD (FEV1 ≤ 50% predicted or modified Medical Research Council (mMRC) dyspnoea scale > 2)
* Patient with severe Chronic Heart Failure (NYHA stage III or IV)
* Patient's refusal of CPAP/APAP treatment support
* Previous CPAP/APAP treatment for Sleep Apnoea
* Patient with ongoing Mandibular Advancement Device (MAD) or in the 12 previous months
* Patient with no permanent place of residence
* Patient participating in another drug or device study within the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
CPAP/APAP adherence evaluation | 3rd month
  average daily number of hours of CPAP/APAP use at 3 months

SECONDARY OUTCOMES:
adherence to CPAP/APAP | 1st, 6th,12th months
  daily average duration of CPAP/APAP use
evolution of daily Apnoea-Hypopnoea Index (AHI) and Non intentional leaks level teletransmitted by CPAP/APAP devices | 1st, 3rd, 6th,12th months
  Daily Apnoea-Hypopnoea Index (AHI) expressed in average daily number per hour and daily non intentional leaks level expressed in L/min as both median and 95th percentile
daytime sleepiness | 1st, 3rd, 6th,12th months
  The numerical answers obtained for the 8 common daily life situations of the Epworth Sleepiness Scale (ESS) are added to calculate the ESS score each time it is collected
Snoring and Quality of Life | 1st, 3rd, 6th,12th months
  The numerical answers obtained for the 5 questions of the snoring questionnaire are added to calculate the snoring score each time the questionnaire is collected. The numerical answer from 0 to 10 obtained on the Quality of Life visual analogue scale is used each time the questionnaire is collected.
For patients in the VitalCare group, Balachandran CPAP perception questionnaire | 1st, 3rd, 6th,12th months
  The numerical answers obtained for the 4 questions regarding difficulty tolerating CPAP, discomfort with CPAP pressure, likelihood of wearing CPAP, and perceived health benefit are added to calculate the CPAP perception score each time it is collected.
Number of contacts between home healthcare provider and patient | 1st, 3rd, 6th,12th months
  The data files extracted from the home healthcare provider database will allow to count for each study patient, the number of contacts between the home healthcare provider and the patient either i) at home, ii) remotely or iii) in care centres
For patients in the VitalCare group, number of updates of the individualised treatment plan | 1st, 3rd, 6th,12th months
  The data files extracted from the home healthcare provider database will allow to count for each patient from the VitalCare group, the number of updates of the individualised treatment plan
adverse events description | through study completion, an average of 1 year
  all adverse events recorded by investigators in the eCRF

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Distrital de Santarém, Santarém, Portugal